CLINICAL TRIAL: NCT05041751
Title: A Pilot Study Assessing the Benefits of Fascial Freedom for the Win (MFR Versus TPI)
Brief Title: Myofascial Release or Trigger Point Injections for the Reduction of Post-Mastectomy Pain Syndrome
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Left Institution
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0498; NCI-2020-13900 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0498 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-03; First posted 2021-09-13 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms | interventions — Acupuncture Points; Massage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm I (trigger point injections) (Active Comparator): Patients receive standard of care trigger point injections at baseline
  Interventions: Procedure: Acupuncture Point Injection; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (myofascial release) (Experimental): Patients perform myofascial release for 10 minutes each day.
  Interventions: Procedure: Massage Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Acupuncture Point Injection — Receive trigger point injections
  Arms: Arm I (trigger point injections)
Procedure: Massage Therapy — Perform myofascial release
  Other Names: Massage
  Arms: Arm II (myofascial release)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies the effect of myofascial release in decreasing post-mastectomy pain compared to standard of care trigger point injections in patients with post-mastectomy pain syndrome. Patients who have mastectomies often experience pain that does not go away after time. This is known as post-mastectomy pain syndrome. Myofascial release is a form of physical therapy in which pressure is applied to the affected areas. Myofascial release may be an effective way of decreasing pain in patients with post-mastectomy pain syndrome without the use of medication.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the change in pain score using the Numerical Rating Scale for pain on an 11-point scale (0-none to 10-worst) from implementation of myofascial release (MFR) versus trigger point injections (TPI) in the treatment of myofascial trigger points (MTP) as noninvasive therapies for post mastectomy pain syndrome (PMPS).

SECONDARY OBJECTIVES:

I. To evaluate the change in medications, particularly opiate medications in the treatment of post mastectomy pain.

II. To evaluate a patient's satisfaction with therapy or treatment throughout the course of the study at each consecutive encounter or follow up.

III. To evaluate a patient's range of motion with therapy or treatment beginning at time of screening and until the end of the study.

IV. To evaluate a patient's degree of lymphedema both subjectively and objectively in the affected extremity(ies) unilateral to the site(s) of mastectomy in response to the various forms of treatment throughout the study.

V. To evaluate quality of life measure changes with treatments used throughout the study.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive standard of care trigger point injections at baseline.

ARM II: Patients perform myofascial release for 10 minutes each day.

ELIGIBILITY:
Inclusion Criteria:

* Chronic post-mastectomy pain syndrome (>= 3 months)
* Able to perform MFR techniques and follow basic instructions
* >= 18 years old

Exclusion Criteria:

* Current chemotherapy
* Pending surgery during treatment
* Active infection
* Active debilitating disease
* Pregnant
* Other chronic pain diagnosis beside PMPS
* Untreated psychiatric diagnosis (not receptive to taking precautions and interventions by treating psychiatrist/psychologist/physician i.e. taking necessary medications)
* Morbid obesity (body mass index [BMI] > 40)
* Allergy history of bupivacaine and/or lidocaine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Pain response | through study completion, an average of 1 year
  Defined by score differences (using the pain numerical rating scale). an 11-point scale (0-none to 10-worst) Pain responders will be defined as patients demonstrating an equal or lower pain score relative to baseline. The 2-week post-treatment assessment will be used to assess the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Le-Short, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org